CLINICAL TRIAL: NCT04846361
Title: The Effectiveness of Vaginal Hygiene Wash as Adjunct Treatment in Bacterial Vaginosis- a Randomized Double Blind Controlled Trial With Microbial Analysis
Brief Title: Vaginal Hygiene Wash as Adjunct Treatment in Bacterial Vaginosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FF-2021-031
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Bacterial Vaginoses
Keywords: vaginal hygiene wash; bacterial vaginosis; microbial analysis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Intervention Model Description: hygiene wash plus antibiotic, placebo wash plus antibiotic
Who Masked: Participant, Investigator
Masking Description: the trial hygiene wash and placebo wash are labelled A or B in identical packaging by manufacturer's company and blinded from both participants and investigators and only revealed at the end of data completion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hygiene wash plus metronidazole (Experimental): Hygiene wash once daily at night for two weeks plus oral metronidazole 400mg three times daily for 1 week
  Interventions: Other: Vaginal hygiene wash
- placebo wash plus metronidazole (Placebo Comparator): Placebo wash once daily at night for two weeks plus oral metronidazole 400mg three times daily for 1 week
  Interventions: Other: placebo wash
- Healthy control (No Intervention): Asymptomatic healthy women with BV negative test

INTERVENTIONS:
Other: Vaginal hygiene wash — vaginal hygiene wash containing Propylene Glycol, Ethylhexylglycerin, Lactic Acid, Sodium Pyrrolidone Carboxylic Acid, Alpha-Glucan Oligosaccharide, Lactococcus Ferment Lysate, Octenidine Hydrochloride plus all other ingredients in placebo wash
  Arms: Hygiene wash plus metronidazole
Other: placebo wash — placebo wash containing water, disodium cocoamphodiacetate, sodium chloride, sodium glycolate, acrylates copolymer, potassium laureate phosphate, tripotassium phosphate, laurel glucoside, lauramidopropyl hydroxysultaine, disulfonate de sodium, Polyethylene glycol (PEG)-120 Methyl Glucose Trioleate, Propanediol, Glycol distearate, Laureth-4, Cocamidopropyl betaine, Potassium Lactate, Caprylyl Glycol, Disodium ethylenediaminetetraacetic acid (EDTA), Potassium Hydroxide, and Perfume
  Arms: placebo wash plus metronidazole

SUMMARY:
This study compares the effect of vaginal hygiene wash versus placebo as adjunct treatment with oral metronidazole in treatment of women with bacterial vaginosis

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing the trial hygiene wash against placebo wash as adjunct treatment with oral metronidazole in women with bacterial vaginosis, with microbial analysis of vaginal flora compared to healthy control women

ELIGIBILITY:
Inclusion Criteria:

* 1. premenopausal women who are sexually active 2.willing to use hygiene wash together with prescribed oral antibiotics 3. able to undergo pelvic examination for sampling of vaginal discharge

Exclusion Criteria:

* 1. Unable to comply with pelvic examination or hygiene wash 2. Concurrent use of hormonal treatment or antibiotic therapy 3. Intrauterine device either copper or levonorgestrel-releasing system 4. Women with known diabetes mellitus 5. Pregnant women

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — non-pregnant women with bacterial vaginosis
Enrollment: 56 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Bacterial vaginosis cure rate | 2 weeks after treatment
  Percentage of participants who have negative bacterial vaginosis (BV) blue test after completed treatment
Visual analog scale of symptoms before treatment | before treatment
  self-evaluation of symptom using Visual analog scale (VAS) scale 0 to 10 based on questionnaire, 5 symptoms assessed are 1) level of comfort in the genital region, 2) malodorous external genitalia, 3) comfort in sexual intercourse, 4) satisfaction regarding intimate hygiene, and 5) self-esteem
Visual analog scale of symptoms after treatment | 2 weeks after treatment
  self-evaluation of symptom using Visual analog scale (VAS) scale 0 to 10 based on questionnaire, 5 symptoms assessed are 1) level of comfort in the genital region, 2) malodorous external genitalia, 3) comfort in sexual intercourse, 4) satisfaction regarding intimate hygiene, and 5) self-esteem
Microbial profile of vaginal flora before treatment | Before treatment
  DNA quantitative polymerase chain reaction (qPCR) array analysis of vaginal swab taken before treatment which includes Lactobacillus, Gardnerella, Prevotella, Candida, and Trichomonas vaginalis
Microbial profile of vaginal flora after treatment | 2 weeks after treatment
  DNA quantitative polymerase chain reaction (qPCR) array analysis of vaginal swab taken before treatment which includes Lactobacillus, Gardnerella, Prevotella, Candida, and Trichomonas vaginalis
Cytokines concentration before treatment | before treatment
  Concentration of cytokines (interleukins (IL-6, IL-8, IL-10), tumor necrosis factor (TNF-alpha) all in pg/mL at baseline
Cytokines concentration after treatment | 2 weeks after treatment
  Concentration of cytokines (interleukins (IL-6, IL-8, IL-10), tumor necrosis factor (TNF-alpha) all in pg/ml after completed treatment

SECONDARY OUTCOMES:
Recurrence of symptoms 1 month after completed treatment | 1 month after completed treatment
  Self-rated symptoms using visual analog scale (VAS) scale 0 to 10 based on questionnaire, 5 symptoms assessed are 1) level of comfort in the genital region, 2) malodorous external genitalia, 3) comfort in sexual intercourse, 4) satisfaction regarding intimate hygiene, and 5) self-esteem
Microbial analysis of vaginal flora 1 month after completed treatment | 1 month after completed treatment
  DNA quantitative polymerase chain reaction (qPCR) array analysis of vaginal swab taken before treatment which includes Lactobacillus, Gardnerella, Prevotella, Candida, and Trichomonas vaginalis

CONTACTS AND LOCATIONS:
Overall Officials: Nur Azurah Abdul Ghani, Principal Investigator — The National University of Malaysia

IPD SHARING:
Plan to Share IPD: Yes
clinical data sheet containing demographics, data collection (VAS score of symptoms, BV blue test)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 20 months

REFERENCES:
- [Background] Lamont RF, Sobel JD, Akins RA, Hassan SS, Chaiworapongsa T, Kusanovic JP, Romero R. The vaginal microbiome: new information about genital tract flora using molecular based techniques. BJOG. 2011 Apr;118(5):533-49. doi: 10.1111/j.1471-0528.2010.02840.x. Epub 2011 Jan 20. PMID 21251190
- [Background] Eusaph AZ, Nighat R, Arshad A. Lactacyd FH as an adjuvant therapy for vulvovaginal infections in Pakistani women: FRESH study, a satisfaction survey. J Pak Med Assoc. 2016 May;66(5):521-7. PMID 27183928
- [Background] Bai G, Gajer P, Nandy M, Ma B, Yang H, Sakamoto J, Blanchard MH, Ravel J, Brotman RM. Comparison of storage conditions for human vaginal microbiome studies. PLoS One. 2012;7(5):e36934. doi: 10.1371/journal.pone.0036934. Epub 2012 May 24. PMID 22655031
- [Background] Hallmaier-Wacker LK, Lueert S, Roos C, Knauf S. The impact of storage buffer, DNA extraction method, and polymerase on microbial analysis. Sci Rep. 2018 Apr 19;8(1):6292. doi: 10.1038/s41598-018-24573-y. PMID 29674641
- [Result] Russo R, Edu A, De Seta F. Study on the effects of an oral lactobacilli and lactoferrin complex in women with intermediate vaginal microbiota. Arch Gynecol Obstet. 2018 Jul;298(1):139-145. doi: 10.1007/s00404-018-4771-z. Epub 2018 Apr 10. PMID 29637269
- [Result] Bahamondes MV, Portugal PM, Brolazo EM, Simoes JA, Bahamondes L. Use of a lactic acid plus lactoserum intimate liquid soap for external hygiene in the prevention of bacterial vaginosis recurrence after metronidazole oral treatment. Rev Assoc Med Bras (1992). 2011 Jul-Aug;57(4):415-20. doi: 10.1590/s0104-42302011000400015. PMID 21876923